CLINICAL TRIAL: NCT02699593
Title: Clinical Evaluation of Approved Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: CR-5809
Record Dates: First submitted 2016-03-01; First posted 2016-03-04 (Estimated); Results first posted 2017-06-09 (Actual); Last update posted 2017-07-12 (Actual); Status verified 2017-06

CONDITIONS: Visual Acuity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Test / Control Sequence (Experimental): Subjects will be dispensed the Test Contact Lens to wear for two weeks, to be worn in a daily wear modality, attending a follow-up visit in 12-17 days. At the follow-up visit, subjects will be dispensed the Control Contact Lens to wear for two weeks, to be worn in a daily wear modality.
  Interventions: Device: Test Contact Lens; Device: Control Contact Lens
- Control / Test Sequence (Active Comparator): Subjects will be dispensed the Control Contact Lens to wear for two weeks, to be worn in a daily wear modality, attending a follow-up visit in 12-17 days. At the follow-up visit, subjects will be dispensed the Test Contact Lens to wear for two weeks, to be worn in a daily wear modality.
  Interventions: Device: Test Contact Lens; Device: Control Contact Lens

INTERVENTIONS:
Device: Test Contact Lens
  Other Names: senofilcon A made with material from a new supplier
Device: Control Contact Lens
  Other Names: senofilcon A made with material from the current supplier

SUMMARY:
This is a 4-week, randomized, double-masked study where subjects will wear bilaterally test and control lenses in random succession. The objective is to evaluate materials from different suppliers.

ELIGIBILITY:
Inclusion Criteria:

1. The subject must read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form.
2. The subject must appear able and willing to adhere to the instructions set forth in this clinical protocol.
3. The subject must be at least 18 and not more than 70 years of age (including 70).
4. The subject's refractive cylinder must be < 0.75 Diopters (D) in each eye.
5. The subject must have best corrected visual acuity of 20/25 or better in each eye.
6. The subject must be a habitual and adapted wearer of ACUVUE® OASYS® brand contact lens in both eyes (at least 1 month of daily wear).
7. The subject must have normal eyes (i.e., no ocular medications or infections of any type).
8. The subject's required spherical contact lens prescription must be in the range of -1.00 D to -6.00 D in each eye.

Exclusion Criteria:

1. Currently pregnant or lactating (subjects who become pregnant during the study will be discontinued).
2. Any ocular or systemic allergies or diseases that may interfere with contact lens wear.
3. Any systemic disease, autoimmune disease, or use of medication that may interfere with contact lens wear.
4. Entropion, ectropion, extrusions, chalazia, recurrent styes, glaucoma, history of recurrent corneal erosions, aphakia.
5. Any previous, or planned, ocular or interocular surgery (e.g., radial keratotomy, photorefractive keratectomy (PRK), laser-assisted in situ keratomileusis (LASIK), etc.)
6. Any grade 3 or greater slit lamp findings (e.g., edema, corneal neovascularization, corneal staining, tarsal abnormalities, conjunctival injection) on the FDA classification scale, any previous history or signs of a contact lens-related corneal inflammatory event (e.g., past peripheral ulcer or round peripheral scar), or any other ocular abnormality that may contraindicate contact lens wear.
7. Any known hypersensitivity or allergic reaction to OPTI-FREE® PureMoist® Contact Lens Solution.
8. Any ocular infection.
9. Any corneal distortion resulting from previous hard or rigid gas permeable contact lens wear.
10. Monovision or multi-focal contact lens correction.
11. Participation in any contact lens or lens care product clinical trial within 14 days prior to study enrollment.
12. History of binocular vision abnormality or strabismus.
13. Any infectious disease (e.g., hepatitis, tuberculosis) or a contagious immunosuppressive disease (e.g., HIV, by self-report).
14. Suspicion of or recent history of alcohol or substance abuse.
15. History of serious mental illness.
16. History of seizures.
17. Employee of investigational clinic (e.g., Investigator, Coordinator, Technician)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2016-04-01 (Actual); Study Completion 2016-04-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Eye Elements Eyecare, Jacksonville, Florida
  - Golden Vision, Sarasota, Florida
  - Advantage Eyecare Associates, LLC, Neodesha, Kansas
  - Advanced Eyecare, PC, Raytown, Missouri
  - Professional Vision Care, Westerville, Ohio
  - Timothy R. Poling, OD, Roanoke, Virginia

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 142 subjects were enrolled into this study. Of the enrolled 1 subject did not meet the eligibility criteria and 141 were dispensed a study lens. Of the dispensed subjects 125 completed the study and 16 subjects were discontinued.
Groups:
- Senofilcon A(Test)/Senofilcon A(Control): Subjects that were randomized to receive the test lens senofilcon A lens first and then the control lens senofilcon A lens second.
- Senofilcon A(Control)/Senofilcon A(Test): Subjects that were randomized to receive the control lens senofilcon A first and then the test lens senofilcon A lens second.
Period: Period 1
Arm/Group | Senofilcon A(Test)/Senofilcon A(Control) | Senofilcon A(Control)/Senofilcon A(Test)
Started | 72 | 69
Completed | 67 | 62
Not Completed | 5 | 7
Not completed — Unsatisfactory Visual Response | 0 | 1
Not completed — Torn Contact Len | 4 | 3
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Adverse Event | 1 | 1
Period: Period 2
Arm/Group | Senofilcon A(Test)/Senofilcon A(Control) | Senofilcon A(Control)/Senofilcon A(Test)
Started | 67 | 62
Completed | 65 | 60
Not Completed | 2 | 2
Not completed — Adverse Event | 1 | 1
Not completed — Lost Contact Lens | 0 | 1
Not completed — Torn Contact Lens | 1 | 0

BASELINE CHARACTERISTICS:
Population: All subjects that were dispensed at least 1 study lens.
Groups:
- Dispensed Subjects: All subjects that were dispensed at least one study lens.
Arm/Group | Dispensed Subjects
Number analyzed (Participants) | 141
Age, Continuous [Mean (Standard Deviation); unit: Years] | 31.0 (8.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 98
  Male | 43
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 11
  Black or African American | 17
  Native Hawaiian or Pacific Islander | 1
  White | 111
  Other | 1
Region of Enrollment [Number; unit: Participants]
  North America | 141

OUTCOME MEASURES:

1. Primary Outcome: Contact Lens Wearing Time
Description: Contact lens wearing time was collected for each subject at the 2-week follow-up evaluation. The average contact lens wearing time in hours was reported for each lens.
Time Frame: 2-week follow-up
Population: Subjects that completed all study visits without a major protocol deviation.
Measure: Mean (Standard Deviation); unit: Hours
Groups:
- Senofilcon A (Test): Subjects that wore the test lens senofilcon A during either the first or second period of the study.
- Senofilcon A (Control): Subjects that wore the control lens senofilcon A lens during the first or second period of the study.
Arm/Group | Senofilcon A (Test) | Senofilcon A (Control)
Number analyzed (Participants) | 118 | 118
Hours | 14.55 (1.534) | 14.63 (1.516)

2. Primary Outcome: Visual Acuity (LogMAR)
Description: Distance Visual Acuity (LogMAR) was assessed using an ETDRS chart at the 2-week follow-up for each subject and eye for 2 conditions, Bright low contrast and Dim high contrast. The average visual acuity (LogMAR) for each condition and lens was reported.
Time Frame: 2-week Follow-up
Population: Subjects that completed all study visits without a major protocol deviation.
Measure: Mean (Standard Deviation); unit: LogMAR
Units Other Than Participants: Eyes
Arm/Group | Senofilcon A (Test) | Senofilcon A (Control)
Number analyzed (Participants) | 118 | 118
Number analyzed (Eyes) | 236 | 236
LogMAR
  Bright Low Contrast | 0.121 (0.0905) | 0.122 (0.0881)
  Dim High Contrast | 0.086 (0.0874) | 0.089 (0.0846)

ADVERSE EVENTS:
Time Frame: Throughout the duration of the study. Approximately 6 weeks per subject.
Arm/Group | Senofilcon A (Test) | Senofilcon A (Control)
Serious Adverse Events (participants affected / at risk) | 0/141 | 0/141
Other Adverse Events (participants affected / at risk) | 0/141 | 0/141

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days